CLINICAL TRIAL: NCT01819181
Title: Women's INternational Transcatheter Aortic Valve Implantation Registry
Acronym: WINTAVI
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Society for Cardiovascular Angiography and Interventions (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 14-1774
Record Dates: First submitted 2013-03-22; First posted 2013-03-27 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Symptomatic Aortic Stenosis
Keywords: TAVI; women; aortic stenosis; VARC2
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study will evaluate all female patients with severe aortic stenosis undergoing transcatheter valve implantation with commercially available valves and delivery systems.

DETAILED DESCRIPTION:
WINTAVI is an international, multi-centre, prospective, observational registry. The purpose of this study is to collect 'real-world' data regarding the clinical utility of all commercially available Transcatheter Aortic Valve Implantation (TAVI) devices for percutaneous aortic valve implantation in female patients with severe Aortic Stenosis (AS) requiring treatment. Data collected in this study will provide additional information on the understanding of the safety and device performance in a 'real-world' setting and how to best treat patients with severe AS. This will include Quality of Life questionnaires (KCCQ).

ELIGIBILITY:
Inclusion Criteria:

1. Severe AS determined by echocardiogram and Doppler, defined as: mean gradient >40 mmHg or peak jet velocity >4.0 m/s and an aortic valve area ≤0.8 cm2 or aortic valve area index ≤0.5 cm2/m2
2. Symptomatic AS demonstrated by angina, congestive heart failure, NYHA functional class ≥ II, or syncope
3. Logistic EuroSCORE suitable for TAVI
4. Patient must have other conditions (such as severe airways disease, porcelain aorta, previous thoracic radiotherapy, Childs Pugh class B and C liver disease) such that the multi-disciplinary team (interventional cardiologists, cardiothoracic surgeons and cardiac anaesthesiologists) agree that co-morbidities render SAVR of high or prohibitive risk.
5. Patient has been informed of the nature of the registry and has provided full written informed consent according to hospital practise

Exclusion Criteria:

1. Patient is not an eligible candidate for TAVI
2. Untreated clinically significant (> 70% obstruction) coronary artery disease in the proximal segments of main branches suitable for revascularization
3. Echocardiographic evidence of intra-cardiac mass, thrombus or vegetation
4. Hemodynamic instability (e.g. requiring inotropic support)
5. Active endocarditis or sepsis within 6-months prior to the study procedure
6. Use of investigational device without CE mark

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive female patients with severe symptomatic Aortic Stenosis who are deemed eligible for TAVI by a multi-disciplinary team in participating sites according to local policy.
Sampling Method: Non-Probability Sample
Enrollment: 1019 (Actual)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
VARC 2 | 30 days
  The primary study endpoint is the VARC 2 early safety endpoint at 30-days (all-cause mortality, all stroke [disabling and non disabling], life-threatening bleeding, stage 2 or 3 acute kidney injury [AKI], coronary artery obstruction requiring intervention, major vascular complications, repeat procedure for valve-related dysfunction).

SECONDARY OUTCOMES:
VARC 2 | up to 2 years
  The clinical efficacy endpoint after 30-days (all-cause mortality, all stroke [disabling and non-disabling], requiring hospitalizations for valve related symptoms or worsening congestive heart failure, NYHA class III or IV, prosthetic valve dysfunction).
BARC | up to 2 years
  Additional individual safety endpoints include the following: all-cause mortality (procedural and 30-days), cardiovascular mortality, MI (peri-procedural and spontaneous), stroke (disabling and non-disabling), bleeding (life-threatening or disabling and major) and BARC type 3a-c and type 5a-b, AKI (stages 2 and 3), incidence of contrast-induced nephropathy, vascular complications (major and minor) and percutaneous closure device failure.
NYHA | up to 2 years
  The New York Heart Association (NYHA) Functional Classification provides a simple way of classifying heart disease (originally cardiac failure), useful for preoperative assessment. It places patients in one of four categories, based on how much they are limited during physical activity:
  Class I: patients with no limitation of activities; they suffer no symptoms from ordinary activities.
  Class II: patients with slight, mild limitation of activity; they are comfortable with rest or with mild exertion.
  Class III: patients with marked limitation of activity; they are comfortable only at rest.
  Class IV: patients who should be at complete rest, confined to bed or chair; any physical activity brings on discomfort and symptoms occur at rest.
KCCQ-12 | up to 2 years
  Kansas City Cardiomyopathy Questionnaire(KCCQ) - a shortened 12 question version of the 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Alaide Chieffo, MD, Principal Investigator — IRCCSSRaffaele and WINSCAI; Roxana Mehran, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (10):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States
- Hôpital Privé Parly 2, Le Chesnay, France
- Italy (4):
  - Azienda Ospedaliero - Ferrarotto Alessi, Catania
  - Instituto Clinico Humanitas, Milan
  - San Raffaele Hospital, Milan
  - Department cardiovascular Sciences Policlinico Umberto I, Rome
- Netherlands (2):
  - Radboud University Nijmegen Medical Center, Nijmegen
  - Erasmus Medical Center Rotterdam, Rotterdam
- Hospital Universitario Miguel Servet, Zaragoza, Spain
- Imperial College, London, United Kingdom

REFERENCES:
- [Background] Buchanan GL, Chieffo A, Montorfano M, Maisano F, Latib A, Godino C, Cioni M, Gullace MA, Franco A, Gerli C, Alfieri O, Colombo A. The role of sex on VARC outcomes following transcatheter aortic valve implantation with both Edwards SAPIEN and Medtronic CoreValve ReValving System(R) devices: the Milan registry. EuroIntervention. 2011 Sep;7(5):556-63. doi: 10.4244/EIJV7I5A91. PMID 21930459
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB; Valve Academic Research Consortium-2. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document. J Thorac Cardiovasc Surg. 2013 Jan;145(1):6-23. doi: 10.1016/j.jtcvs.2012.09.002. Epub 2012 Oct 16. PMID 23084102
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Hayashida K, Morice MC, Chevalier B, Hovasse T, Romano M, Garot P, Farge A, Donzeau-Gouge P, Bouvier E, Cormier B, Lefevre T. Sex-related differences in clinical presentation and outcome of transcatheter aortic valve implantation for severe aortic stenosis. J Am Coll Cardiol. 2012 Feb 7;59(6):566-71. doi: 10.1016/j.jacc.2011.10.877. PMID 22300690
- See also: Women in Innovations ("WIN") mission is to address sex-based disparities in cardiovascular diagnosis, treatment and outcomes through innovative educational and research activities. — http://www.scai.org/win